CLINICAL TRIAL: NCT01890486
Title: The Prospective Collection, Storage and Reporting of Data on Patients
Brief Title: The Prospective Collection, Storage and Reporting of Data on Patients Undergoing Hematopoietic Stem Cell Transplantation Utilizing a Standard Preparative Regimen
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CCCWFU 95300
Record Dates: First submitted 2013-06-27; First posted 2013-07-01 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Non-Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma; Germ Cell Neoplasms; Myelodysplastic Syndromes; Chronic Lymphocytic Leukemia; Immunodeficiency Diseases
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Neoplasms, Germ Cell and Embryonal; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To provide the IRB approved mechanism for the prospective collection, analysis and reporting of data on patients who are undergoing either an autologous or allogeneic hematopoietic stem cell transplant for a disease in which a research question is not being addressed and for which peer reviewed, published data have demonstrated efficacy for this treatment approach.

ELIGIBILITY:
Inclusion Criteria:

Planned standard of care dose intensive therapy and either an allogeneic or autologous bone marrow transplant

Exclusion Criteria:

Participation in any other treatment research protocol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are not on a specific "treatment research protocol" but who are nevertheless receiving "standard of care" dose intensive therapy and either an allogeneic or autologous bone marrow transplant
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2001-05-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Data followup | 1 year
  Gather basic survival and complication data for operational and research databases for ongoing regulatory and future operational queries

CONTACTS AND LOCATIONS:
Overall Officials: Dianna Howard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States